CLINICAL TRIAL: NCT02605356
Title: A Phase 1b/2 Trial to Evaluate the Safety and Efficacy of Radium-223 Dichloride (BAY88-8223) in Combination With Bortezomib and Dexamethasone in Early Relapsed Multiple Myeloma
Brief Title: Phase 1b/2 Study Testing Radium-223 Dichloride/Bortezomib/Dexamethasone Combination in Relapsed Multiple Myeloma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study restarted under new study number 18987
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17451; 2015-000427-82 (EudraCT Number)
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-09

CONDITIONS: Multiple Myeloma
Keywords: Radium-223 dichloride; bortezomib; dexamethasone; early relapsed multiple myeloma; combination therapy multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — radium Ra 223 dichloride; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Radium-223 dichloride [Phase 1, dose 1] (Experimental): Phase 1: Radium-223 dichloride; 30 kiloBecquerel (kBq)/kg body weight (33 kBq/kg after implementation of National Institute of Standards and Technology [NIST] update) every 4 weeks for a total of 6 radium-223 dichloride doses plus SOC bortezomib/dexamethasone.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Bortezomib; Drug: Dexamethasone
- Radium-223 dichloride [Phase 1, dose 2] (Experimental): Phase 1: Radium-223 dichloride; 50 kBq/kg body weight (55 kBq/kg after implementation of NIST update) every 4 weeks for a total of 6 radium-223 dichloride doses plus SOC bortezomib/dexamethasone.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Bortezomib; Drug: Dexamethasone
- Radium-223 dichloride [Phase 1, dose 3] (Experimental): Phase 1: Radium-223 dichloride; 80 kBq/kg body weight (88 kBq/kg after implementation of NIST update) every 4 weeks for a total of 6 radium-223 dichloride doses plus SOC bortezomib/dexamethasone.
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Bortezomib; Drug: Dexamethasone
- Placebo +SoC [Phase 2] (Placebo Comparator): Phase 2: Matching placebo (isotonic saline) every 4 weeks for a total of 6 doses plus SoC (Standard of care) bortezomib/dexamethasone.
  Interventions: Drug: Placebo; Drug: Bortezomib; Drug: Dexamethasone
- Radium-223 dichloride + SoC [Phase 2] (Experimental): Phase 2: Phase 1b-selected dose of radium-223 dichloride every 4 weeks for 6 doses plus SOC bortezomib/dexamethasone
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223)
  Arms: Radium-223 dichloride + SoC [Phase 2]; Radium-223 dichloride [Phase 1, dose 1]; Radium-223 dichloride [Phase 1, dose 2]; Radium-223 dichloride [Phase 1, dose 3]
Drug: Placebo
  Arms: Placebo +SoC [Phase 2]
Drug: Bortezomib
Drug: Dexamethasone

SUMMARY:
This study will be conducted in 2 parts. The phase 1b part will be an international, phase 1b, open-label, dose-escalation assessment of radium-223 dichloride administered with bortezomib and dexamethasone in subjects with relapsed multiple myeloma. The primary endpoint of the phase 1b part is to determine the optimal dose of radium-223 dichloride in combination with bortezomib/dexamethasone for the Phase 2 portion of the study.

The phase 2 part will be an international, phase 2, double-blind, randomized, placebo-controlled assessment of radium-223 dichloride versus placebo administered with bortezomib and dexamethasone, in subjects with relapsed multiple myeloma. Randomization (1:1) in the phase 2 part will be stratified by:

* Prior bortezomib treatment (yes, no)
* Prior treatment (1 prior line of treatment, >1 prior line of treatment) Approximately 30 subjects (10 subjects per cohort) will be enrolled in the phase 1b part of the study and approximately 196 subjects will be enrolled in the phase 2 part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed diagnosis of multiple myeloma
* Subjects must have received at least 1 and not more than 3 previous lines of treatment and have had a response to treatment (i.e., achieved a minimal response [MR] or better) according to the International Myeloma Working Group (IMWG) uniform response criteria
* Subjects must have had progressive disease according to the IMWG uniform response criteria following the last multiple myeloma treatment
* Subjects must have measurable disease defined as at least 1 of the following (according to central laboratory results):

  * Serum M-protein ≥1 g/dL
  * Urine M-protein ≥200 mg/24 hours
  * Serum free light chain (FLC) ≥10 mg/dL with abnormal ratio
* ≥1 bone lesion identifiable by radiograph, computed tomography, magnetic resonance imaging, or bone scintigraphy
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2
* Subjects must be nonrefractory to bortezomib and had no progression during or within 60 days after completion of bortezomib
* Absolute neutrophil count (ANC) ≥1.5 × 10e9/L, hemoglobin (Hb) ≥9.0 g/dL, and platelet count ≥75.0 × 10e9/L independent of transfusion of red blood cells (RBC) or platelet concentrates and independent of granulocyte colony stimulating factor (G-CSF) or granulocyte macrophage colony stimulating factor (GM-CSF)

Exclusion Criteria:

* Systemic glucocorticoid therapy (prednisone >10 mg/day orally or equivalent) within the last 4 weeks prior to first dose, unless tapered and on a stable dose ≤10 mg/day for at least 1 week
* Subjects with known POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or light chain (AL) amyloidosis
* Plasma cell leukemia
* Systemic anti-cancer therapy within 4 weeks prior to first dose
* Radiation therapy in the previous 4 weeks prior to first dose except if given for pain management and involves less than 10% of the bone marrow
* Prior treatment with radium-223 dichloride or any experimental radiopharmaceutical
* Congestive heart failure (New York Heart Association [NYHA] class III to IV), symptomatic cardiac ischemia, cardiomyopathy, clinically relevant ventricular arrhythmia, pericardial disease, unstable angina or myocardial infarct in the previous 6 months prior to first dose, left ventricular ejection fraction <40%
* Neuropathy ≥ Grade 2 or Grade 1 with pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2019-11 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Joint positive adjudication of safety summary in Phase 1b by steering committee, investigator and sponsor (Yes/No) | At 13 months
Progression-free survival (PFS) in Phase 2, defined as the time (in days) from date of randomization to disease progression | Up to 25 months

SECONDARY OUTCOMES:
Objective response rate (ORR) in Phase 1b, in the proportion of subjects in the analysis population who have complete response (CR), stringent complete response (sCR), very good partial response (VGPR), partial response (PR), or stable disease (SD) | Approximately 12 months
Duration of response in Phase 1b, defined as the time (in days) from the date of first response to treatment (CR, sCR, VGPR, PR) to the date of disease progression or death | Approximately 12 months
Number of participants with adverse events in phase 2 | Up to 25 months
Overall survival (OS) in Phase 2, defined as the time (in days) from date of randomization until death from any cause | Up to 25 months
Time to Symptomatic Skeletal Event (SSE) in Phase 2, defined as the time (days) from the date of randomization to the date of the first on-study SSE | Up to 25 months
Symptomatic skeletal event free survival in Phase 2, defined as the time from randomization to the occurrence of 1 of the following: First on-study SSE or Death from any cause if death occurs before a documented SSE | Up to 25 months
Time to pain progression in Phase 2 | Up to 25 months
Duration of response in Phase 2 | Up to 25 months
Objective Response Rate (ORR) in Phase 2 | Up to 25 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (51):
- United States (10):
  - Scottsdale, Arizona
  - Little Rock, Arkansas
  - Encinitas, California
  - Metairie, Louisiana
  - Rockville, Maryland
  - New York, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Watertown, South Dakota
  - Seattle, Washington
- Australia (2):
  - Adelaide, South Australia
  - Box Hill
- Belgium (4):
  - Bruges
  - Bruxelles - Brussel
  - Liège
  - Yvoir
- Québec, Quebec, Canada
- Germany (4):
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Mainz, Rhineland-Palatinate
  - Berlin, State of Berlin
- Greece (2):
  - Athens
  - Rio / Patra
- Israel (5):
  - Afula
  - Haifa
  - Jerusalem
  - Ramat Gan
  - Ẕerifin
- Italy (8):
  - Bologna, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Milan, Lombardy
  - Novara, Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Florence, Tuscany
  - Pisa, Tuscany
- South Korea (4):
  - Goyang-si, Gyeonggido
  - Daegu
  - Jeollanam-do
  - Seoul
- Spain (8):
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - San Sebastián, Guipúzcoa
  - Palma de Mallorca, Illes Baleares
  - Madrid, Madrid
  - Seville, Sevilla
  - Valencia, Valencia
  - Barcelona
- Taiwan (3):
  - Taipei, Taipei
  - Taichung
  - Taipei